CLINICAL TRIAL: NCT00824460
Title: An Open-label, Randomised, Active Controlled Multi-center Phase II Dose Finding Study to Evaluate the Ability of PA21 to Lower Serum Phosphate Levels and the Tolerability in Patients With Chronic Kidney Disease on Maintenance Hemodialysis
Brief Title: Study of Phosphate Levels in Patients With Chronic Kidney Disease
Acronym: PA21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA-CL-03A; 75610
Record Dates: First submitted 2009-01-09; First posted 2009-01-16 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Iron; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1.25 g PA21 (Experimental)
  Interventions: Drug: 1.25 g PA21 (250 mg iron)
- 5.0 g PA21 (Experimental)
  Interventions: Drug: 5.0 g PA21 (1,000 mg iron)
- 7.5 g PA21 (Experimental)
  Interventions: Drug: 7.5 g PA21 (1,500 mg iron)
- 10.0 g PA21 (Experimental)
  Interventions: Drug: 10.0 g PA21 (2,000 mg iron)
- 12.5 g PA21 (Experimental)
  Interventions: Drug: 12.5 g PA21 (2,500 mg iron)
- Sevelamer hydrochloride - active control (Experimental)
  Interventions: Drug: Sevelamer hydrochloride

INTERVENTIONS:
Drug: 1.25 g PA21 (250 mg iron) — Daily dose of 1.25 g PA21 (1 tablet/day) for 6 weeks. One PA21 tablet will be taken orally with the largest meal of the day.
  Arms: 1.25 g PA21
Drug: 5.0 g PA21 (1,000 mg iron) — Daily dose of 5.0 g PA21 (4 tablets/day) for 6 weeks. Two PA21 tablets will be taken orally with the largest meal of the day, and one PA21 tablet will be taken orally with each of the two smaller main meals of the day (3 meals per day).
  Arms: 5.0 g PA21
Drug: 7.5 g PA21 (1,500 mg iron) — Daily dose of 7.5 g PA21 (6 tablets/day) for 6 weeks. Two PA21 tablets will be taken orally with each of the three main meals of the day (3 meals per day).
  Arms: 7.5 g PA21
Drug: 10.0 g PA21 (2,000 mg iron) — Daily dose of 10.0 g PA21 (8 tablets/day) for 6 weeks. Four PA21 tablets will be taken orally with the largest meal of the day, and two PA21 tablets will be taken orally with each of the two smaller main meals of the day (3 meals per day).
  Arms: 10.0 g PA21
Drug: 12.5 g PA21 (2,500 mg iron) — Daily dose of 12.5 g PA21 (10 tablets/day) for 6 weeks. Four tablets will be taken orally with the largest meal of the day, and three PA21 tablets will be taken orally with each of the two smaller main meals of the day (3 meals per day).
  Arms: 12.5 g PA21
Drug: Sevelamer hydrochloride — Daily dose of 4.8 g Sevelamer hydrochloride (6 tablets/day) for 6 weeks. Two Sevelamer tablets will be taken orally with each of the three main meals of the day (3 meals per day).
  Arms: Sevelamer hydrochloride - active control

SUMMARY:
The purpose of this study is to investigate the ability of different doses of PA21 to lower serum phosphate levels, in patients with chronic kidney disease on maintenance hemodialysis.

ELIGIBILITY:
Main Inclusion Criteria:

* ≥ 18 years of age,
* Receiving stable maintenance hemodialysis 3 times a week
* On restricted phosphate diet at screening and throughout study
* Receiving stable dose of phosphate binder for at least 1 month
* Serum phosphate levels >1.78 mmol/L

Main Exclusion Criteria:

* Uncontrolled hyperphosphatemia
* Hypercalcemia at screening or during washout
* Serum calcium < 1.9 mmol/L (<7.6 mg/dL)
* Severe hyperparathyroidism (iPTH levels >600 ng/L)
* Pregnancy or lactation
* Iron deficiency anemia
* History of hemochromatosis or ferritin >800 mg/L,
* Hepatitis B, hepatitis C or other significant concurrent liver disorders
* Known positivity to HIV
* Use of oral iron preparations 1 month before screening,
* Serious medical condition or uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rudolf P Wutrich, MD, Principal Investigator — Unafilliated
Locations (59):
- United States (9):
  - Western Nephrology & Metabolic Disease, Arvada, Colorado
  - Complete Renal Care, Denver, Colorado
  - Pines Clinical Research, Pembroke Pines, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Nephrology Associates, Fresh Meadows, New York
  - University Hospitals / Case Medical Center, Cleveland, Ohio
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Nephrology Associates, Nashville, Tennessee
  - Southwest Houston Research, Houston, Texas
- Bulgaria (10):
  - MHAT, Gabrovo
  - MHAT Plovdiv, Plovdiv
  - Department of Haemodialysis at MHAT, Rousse
  - 5th MHAT Sofia, Sofia
  - SHATCVD - National Cardiology Hospital, Sofia
  - MHAT "Tokuda Hospital Sofia", Sofia
  - UMHAT "Alexandrovska" Dialysis Clinic, Sofia
  - UMHAT "Sveti Ivan Rilski", Sofia
  - UMHAT "Sveta Anna", Sofia
  - MDHAT Department of Haemodialysis and Nephrology, Veliko Tarnovo
- Croatia (10):
  - Opca bonica Bjelovar, Bjelovar
  - Opca bolnica Karlovac, Karlovac
  - Opca bolnica, Koprivnica
  - Klinicka bolnica Osijek, Osijek
  - Klinicki bolnicki centar Rijeka, Rijeka
  - Klinicki bolnicki centar Split, Split
  - Opca bolnica Zadar, Zadar
  - Klinicka bolnica, Zagreb
  - Poliklinika Sveti Duh II, Zagreb
  - Klinicka bolnica Dubrava, Zagreb
- Czechia (4):
  - Innef a.s. Hemodialyzancni stredisko, Brno
  - Nemocnice Nove Mesto na Morave, Nove Město Na Morave
  - Nemocnice s poliklinikou v Novem Jicine, Nový Jičín
  - Klinika nefrologie VFN, Prague
- Germany (2):
  - Nephrologische Gemeinschaftspraxis und Dialysezentrum, Dortmund
  - Marienhospital, Herne
- Poland (7):
  - Niepubliczny Zaklad Opieki Zdrowotnej, Golub-Dobrzyń
  - Katedra i Klinika Nefrologii, Katowice
  - NZOZ Dializa, Olkusz
  - Katedra i Klinika Nefrologii, Poznan
  - Samodzielny Specjalistyczny, Siedlce
  - Niepubliczny Zaklad Opieki Zdrowotnej, Sieradz
  - Centrum Dializy i Diagnostyki, Warsaw
- Romania (5):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic, Lasi
  - SC Renamed Nefrodial SRL, Oradea
  - S.C. Avitum S.R.L, Târgu Mureş
- Russia (9):
  - GOU VPO Kazan, Kazan'
  - GUZ City Clinical Hospital, Moscow
  - MUZ City Clinical Hospital, Novosibirsk
  - Saint-Petersburg CUS City Mariinskaya Hospital, Saint Petersburg
  - Saint-Petersburg GUZ City Clinical Hospital, Saint Petersburg
  - GOU VPO, Saint Petersburg
  - Saint-Petersburg GUZ City Hospital, Saint Petersburg
  - CUS City Hospital, Saint Petersburg
  - MLPU Clinical City Hospital, Smolensk
- Switzerland (3):
  - Kantonspital Aarau, Aarau
  - Chuv Lausanne, Lausanne
  - Universitatsspital Zurich, Zurich

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.25 g PA21 (250 mg Iron): Daily dose of 1.25 g PA21 (1 tablet)
- 5.0 g PA21 (1,000 mg Iron): Daily dose of 5.0 g PA21 (4 tablets)
- 7.5 g PA21 (1,500 mg Iron): Daily dose of 7.5 g PA21 (6 tablets)
- 10.0 g PA21 (2,000 mg Iron): Daily dose of 10.0 g PA21 (8 tablets)
- 12.5 g PA21 (2,500 mg Iron): Daily dose of 12.5 g PA21 (10 tablets)
- Sevelamer Hydrochloride - Active Control: Daily dose of 4.8 g Sevelamer hydrochloride (6 tablets)
Period: Overall Study
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0 g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5 g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control
Started | 26 | 26 | 25 | 27 | 24 | 26
Completed | 18 | 17 | 20 | 15 | 15 | 18
Not Completed | 8 | 9 | 5 | 12 | 9 | 8

BASELINE CHARACTERISTICS:
Population: For baseline characteristics data, from All Randomised patients was used.
Groups:
- 10.0 g PA21 (2,000 mg Iron): Daily dose of 10.0g PA21 (8 tablets)
- 12.5g PA21 (2,500 mg Iron): Daily dose of 12.5 g PA21 (10 tablets)
- Total: Total of all reporting groups
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0 g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control | Total
Number analyzed (Participants) | 26 | 26 | 25 | 27 | 24 | 26 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 14 | 17 | 14 | 16 | 93
  >=65 years | 12 | 8 | 11 | 10 | 10 | 10 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.29) | 59.7 (13.80) | 61.9 (13.71) | 60.6 (12.74) | 59.3 (12.32) | 61.1 (11.00) | 60.5 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 9 | 10 | 11 | 11 | 57
  Male | 17 | 19 | 16 | 17 | 13 | 15 | 97
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 3 | 4 | 2 | 4 | 21
  Czech Republic | 0 | 3 | 0 | 0 | 3 | 2 | 8
  Poland | 4 | 2 | 3 | 2 | 0 | 4 | 15
  Romania | 2 | 4 | 2 | 3 | 1 | 0 | 12
  Croatia | 5 | 3 | 9 | 8 | 8 | 7 | 40
  Russian Federation | 7 | 5 | 3 | 5 | 2 | 6 | 28
  Bulgaria | 3 | 3 | 5 | 4 | 7 | 1 | 23
  Germany | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Switzerland | 0 | 2 | 0 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum-phosphate Levels at the End of Treatment.
Time Frame: 6 weeks after baseline
Population: For the Primary Outcome, data from the Full Analysis Set (FAS) was used. The FAS consists of all randomised subjects who received at least 1 dose of study treatment and had at least 1 post-baseline efficacy evaluation (while on treatment).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0 g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control
Number analyzed (Participants) | 26 | 26 | 25 | 25 | 24 | 24
mmol/L | -0.042 (0.650) | -0.348 (0.684) | -0.404 (0.391) | -0.644 (0.551) | -0.547 (0.584) | -0.341 (0.436)

2. Secondary Outcome: Change From Baseline in Serum-phosphate Levels at Week 2
Time Frame: 2 weeks after baseline
Population: For this Secondary Outcome, FAS was used, which consists of all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline efficacy evaluation (while on treatment).
  Number of participants analyzed at this time point includes all subjects that had serum-phosphate measured at Week 2.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0 g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5 g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control
Number analyzed (Participants) | 26 | 26 | 25 | 24 | 24 | 24
mmol/L | -0.03 (0.55) | -0.36 (0.35) | -0.41 (0.40) | -0.47 (0.62) | -0.46 (0.45) | -0.41 (0.44)

3. Secondary Outcome: Change From Baseline in Serum-phosphate Levels at Week 4
Time Frame: 4 weeks after baseline
Population: For this Secondary Outcome, FAS was used, which consists of all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline efficacy evaluation (while on treatment).
  Number of participants analyzed at this time point includes all subjects that had serum-phosphate measured at Week 4.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- 1.25 g PA21 (250 mg Iron): Daily dose of 1.25g PA21 (1 tablet)
- 5.0g PA21 (1,000 mg Iron): Daily dose of 5.0g PA21 (4 tablets)
- 7.5 g PA21 (1,500 mg Iron): Daily dose of 7.5g PA21 (6 tablets)
- 12.5g PA21 (2,500 mg Iron): Daily dose of 12.5g PA21 (10 tablets)
- Sevelamer Hydrochloride - Active Control: Daily dose of 4.8g sevelamer hydrochloride (6 tablets)
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control
Number analyzed (Participants) | 24 | 23 | 22 | 21 | 21 | 22
mmol/L | -0.03 (0.39) | -0.39 (0.45) | -0.32 (0.54) | -0.58 (0.53) | -0.53 (0.48) | -0.53 (0.35)

4. Secondary Outcome: Change From Baseline in Serum-phosphate Levels at Week 5
Time Frame: 5 weeks after baseline
Population: For this Secondary Outcome, FAS population was used, which consists of all randomized subjects who received at least 1 dose of study treatment and had at least 1 post-baseline efficacy evaluation (while on treatment).
  Number of participants analyzed at this time point includes all subjects that had a serum-phosphate measurement at Week 5.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0 g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5 g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control
Number analyzed (Participants) | 24 | 21 | 21 | 19 | 20 | 20
mmol/L | -0.05 (0.62) | -0.51 (0.62) | -0.40 (0.33) | -0.57 (0.55) | -0.58 (0.58) | -0.52 (0.37)

ADVERSE EVENTS:
Description: For the serious adverse event (SAE) and adverse event (AE) listings, data from the Safety Set (SS) was used. The SS consists of all randomised subjects who received at least 1 dose of study treatment.
Arm/Group | 1.25 g PA21 (250 mg Iron) | 5.0 g PA21 (1,000 mg Iron) | 7.5 g PA21 (1,500 mg Iron) | 10.0 g PA21 (2,000 mg Iron) | 12.5 g PA21 (2,500 mg Iron) | Sevelamer Hydrochloride - Active Control
Serious Adverse Events (participants affected / at risk) | 2/26 | 2/26 | 1/25 | 1/27 | 2/24 | 2/26
Other Adverse Events (participants affected / at risk) | 13/26 | 16/26 | 13/25 | 18/27 | 17/24 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.25 g PA21 (250 mg Iron) (N=26) | 5.0 g PA21 (1,000 mg Iron) (N=26) | 7.5 g PA21 (1,500 mg Iron) (N=25) | 10.0 g PA21 (2,000 mg Iron) (N=27) | 12.5 g PA21 (2,500 mg Iron) (N=24) | Sevelamer Hydrochloride - Active Control (N=26)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.25 g PA21 (250 mg Iron) (N=26) | 5.0 g PA21 (1,000 mg Iron) (N=26) | 7.5 g PA21 (1,500 mg Iron) (N=25) | 10.0 g PA21 (2,000 mg Iron) (N=27) | 12.5 g PA21 (2,500 mg Iron) (N=24) | Sevelamer Hydrochloride - Active Control (N=26)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 8 | 7 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 1 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1 | 2
Faeces Discoloure (Gastrointestinal disorders) | 2 | 3 | 3 | 4 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not present or publish partial or complete study results individually. Any manuscript or abstract proposed by the Investigators must be reviewed and approved in writing by Vifor Pharma before submission for publication. Names of all Investigators participating in the study will be included in the publication.